CLINICAL TRIAL: NCT00523172
Title: A Randomized Clinical Trial Comparing Two Manipulative Protocols to Assess Changes in Pain, ROM, Quality of Life, Cost and Risk for Falls in Subjects With Hip Osteoarthritis
Brief Title: Clinical Assessment of Two Manipulative Protocols in Treatment of Hip Osteoarthritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cleveland Chiropractic College (Other)
Collaborators: Durban University of Technology (Other); Macquarie University, Australia (Other)
Responsible Party: James W Brantingham, DC, PhD, Cleveland Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB08102007
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Osteoarthritis, Hip
Keywords: Chiropractic Manipulation
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Musculoskeletal Manipulations; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Active Comparator): 1) Group A will receive 9 manipulative therapy treatments (adjustments) to one area: the hip with pre-manipulative static and post active-assisted stretch of tight hip muscles. After the last (or 9th) treatment these patients will receive general advice and recommendations on managing HOA and how to gently and safely increase general exercise.
  • Based on a previous trial, Group A treatment appears superior than placebo. There will be a 3, 6 and 9 month follow up.
  Interventions: Procedure: manual or manipulative therapy
- Group B (Active Comparator): 2) Group B will receive 9 treatments with manipulative therapy treatments (adjustments) to the entire kinetic chain (five areas): the lumbosacral, sacroiliac, hip, knee, ankle and foot joints with pre-manipulative static and post active-assisted stretch of tight hip muscles. There will be a 3, 6 and 9 month follow up.
  Interventions: Procedure: Manual / Manipulative Therapy
- Supportive Care (Other): Supportive Care 3) Groups A and B will receive supportive care after the 9th visit consisting of (up to a maximum of) 6 visits, PRN or as needed, until the 9 month follow up. This is to see if peak gains may be maintained (as noted in the previous trial) throughout the follow up period.
  Enrolled subjects will commonly receive 2 treatments per week (occasionally, less or more than 1 to 2 treatments per week due to (College or University) semester breaks, exams, clinic closures and so forth) until 9 treatments are completed.
  Interventions: Procedure: Supportive Care

INTERVENTIONS:
Procedure: manual or manipulative therapy — Active comparator will receive 9 treatments of manual or manipulative therapy to the hip (HVLA hip manipulations per protocol 1) with pre-manipulative static and post manipulative active-assisted stretch of hip muscles after each manipulation.
  Arms: Group A
Procedure: Manual / Manipulative Therapy — Active comparator will receive 9 treatments of manual or manipulative therapy to the lumbosacral, sacroiliac, hip and knee, ankle and foot joints (HVLA and Grades I-IV mobilization per protocol 2) stretching and exercise.)
  Arms: Group B
Procedure: Supportive Care — Supportive Care 3) Groups A and B will receive supportive care after the 9th visit consisting of (up to a maximum of) 6 visits, PRN or as needed, until the 9 month follow up. This is to see if peak gains may be maintained (as noted in the previous trial) throughout the follow up period.
  Enrolled subjects will commonly receive 2 treatments per week (occasionally, less or more than 1 to 2 treatments per week due to (College or University) semester breaks, exams, clinic closures and so forth) until 9 treatments are completed.
  Arms: Supportive Care

SUMMARY:
Purpose of this study is to examine the effect of chiropractic adjusting (manipulative therapy) and rehabilitation on hip osteoarthritis (hip OA) in older adults.

DETAILED DESCRIPTION:
Patients seek treatment from chiropractors for (OA). OA is the fifth most reported and treated disorder in medical practice. Osteoarthritis of the hip (OAH), a subset, affects ≥12 million American adults and leads to pain, loss of mobility, decreased: function, strength, activities of daily living, quality of life and is a significant risk factor for falls. Medical care prescribed for OAH is lifestyle accommodation (a cane, high chairs and toilet seats, etc), non-steroidal anti-inflammatory drugs (NSAIDS), anti-arthritics, steroids, various and sundry prescription and non-prescription medications and exercise. Randomized controlled trials (RCTS) support exercise for knee OA (KOA) treatment, proven superior to placebo, less so for OAH. Ninety-two percent of patients with OAH use NSAIDS. Frequent minor and intermittently serious adverse reactions to chronic use of NSAIDS and evidence that manipulative/manual therapy (MAN) and exercise/rehabilitation therapy may give equivalent relief, suggests NSAIDS should be infrequently used. Supported by an earlier RCT that demonstrated manual, soft tissue and exercise therapy for KOA superior to placebo; later this protocol was found superior to exercise. A similar multimodal (multimodal = MAN with 2 or more combined treatments) 2004 RCT compared exercise protocol versus MAN combined with passive and active stretch for OAH. Early, superior relief and function was achieved with multimodal MAN. This suggests multimodal MAN (manipulative) therapy may be a superior treatment.

In studies that followed multimodal MAN over a year (without minimal, later, PRN or supportive treatment given) all treatment benefits begin to decrease toward a similar mean). One feature frequently inherent in previous trial design has no availability of additional brief treatment rounds subsequent to a short course of interventional therapy. Researchers typically design interventions in search of evaluating short-term interventional strategies where sustained improvements in symptom relief, function, and QoL (quality of life) will be achieved. The current investigators question the utility of such an approach. Frequently patients experience minor setbacks in their improvement secondary to minor injuries or diminution in compliance over time with exercise programs. Combining the practical awareness of patient experience during the follow-up interval with the reality of the typically ongoing nature of OA activity has stimulated the need for some reasonable level of and access to follow-up care after the initial treatment course. A patient who has responded to the initial brief intervention course but who subsequently requires an occasional office visit for physical re-evaluation, review of exercise and a visit or two of manual methods is not inherently synonymous with a failed interventional approach any more that repeat doses of pharmaceuticals are required for other chronic conditions whether it be NSAIDs for OA or insulin for diabetes.

Significant morbidity and occasional mortality from NSAID and drug-related complications and surgery; difficulty in obtaining compliance with prolonged exercise protocols; apparent equivalent (manipulative) outcomes (in pain relief, mobility and function); falls with appalling sequela in morbidity, mortality and expense, justifies further research into multimodal manipulative therapy for treatment of OAH. Data suggests such therapy may give earlier, effective, less costly outcomes and reflects a common clinical chiropractic approach to OAH. In addition to the hip joint, OAH disability is significantly worsened by restricted knee flexion; and in a similar vein, KOA is made worse by hip joint stiffness and dysfunction. Manipulative therapy to a fuller, or the full, kinetic chain (lumbosacral through foot) appears superior for Knee and hip OA. The 2nd, new protocol (protocol 2) will be compared to the 1st (or Hoeksma et al like protocol 1). Additional PRN treatment for both protocols is added to maintain or restore peak levels of improvement (see above and below).

Specific Aim 1: Recruit a pool of HOA patients from senior centers, the local community, medical and chiropractic clinics, and through advertising in collaboration with other Universities/Colleges or Schools.

Specific Aim 2: Establish protocols for long-term surveillance of OAH in chiropractic patients. This study will take 2 years. Recruitment will be during the first 9 months. Core measurements and data will be collected: at baseline; blind measurements after the 9th treatment, and 3, 6, and a 9 month follow up. After the end of the 9th treatment(per protocol 2), additional PRN treatment 1-3 visits every 1-3 months up to 6 months (not to exceed 6 additional visits before 9 months after beginning care).

Specific Aim 3: integrate a clinical research program with a teaching clinic system.

Specific Aim 4: Analysis: collect and compare outcome data comparing protocols. Primary outcome measure: The McMaster Overall Therapy Effectiveness (the OTE) Tool for determining general improvement, satisfaction and the importance of changes to, and experienced by, the patient. Secondary outcome measures: WOMAC, Harris Hip Scale, Goniometry, the One Legged Standing test and Berg Balance Scale.

Specific Aim 5: Cost Includes tracking: time, procedures and costs at each visit by CPT codes. CPT data will be analyzed by various means after completion of the trial.

a) Minimum outcome measure: Appropriate CPT codes marked at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Hip pain and < 15° internal rotation and < than 115° flexion or
* Hip pain with >15° internal rotation causing hip pain and morning stiffness ≤ 60 minutes Note: Hip x-rays will be taken in each case (after a clinical diagnosis of hip osteoarthritis has been made and to rule out and exclude severe pathology) to determine grades (0-4) Kellgren Lawrence x-ray scale. If medically necessary, lumbosacral pelvic x-rays will be obtained-- see exclusions below)
* Age ≥ 60 and ≤ 85 years of age
* Diagnosis of concurrent subluxation complex

  * Diagnosis of subluxation complex (aka segmental joint dysfunction) will be supported throughout using the PART(S) system.
* Additionally, OAH patients, who demonstrate a + One Legged Standing Test (OLST) and + Berg Balance Scale (BBS) will be monitored as a subgroup (with OLST and BBS) at all assessments.

Exclusion Criteria:

General and internal medical disorders such as:

* Significant visual disorders
* Severe vestibular disorders (i.e., Meniere's)
* Neurological (including Alzheimer's and other degenerative brain and mental disorders, disease and dysfunction) peripheral sensory disorders (severe insulin dependent diabetes)
* Hip joint replacement
* RA
* Instability
* Fracture/ and severe osteoporosis
* Frank avascular necrosis with or without moderate or severe deformity
* Lumbar herniated disc and injury
* Severe balance and proprioception problems (i.e., inability to stand with and/or without marked spinal or hip deformity) etc.
* Symptoms (moderate to severe) in both hips.
* Marked or severe fear of chiropractic adjustments/manipulative and or exercise procedures.
* Breaks for treatment longer than 3-4 weeks depending on each circumstance or merit may be construed as non-compliance and may be excluded.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Recruit a pool of HOA patients from senior centers, the local community, medical and chiropractic clinics, and through advertising in collaboration with other Universities/Colleges or Schools. | Nine Months
Establish protocols for long-term surveillance of OAH in chiropractic patients. | 2 years
integrate a clinical research program with a teaching clinic system. | Two years
Collect and compare protocol outcome data. Primary outcome measure will be: a 6 point Likert scale. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Brantingham, D.C., Ph.D., Principal Investigator — Cleveland Chiropractic College
Locations (3):
- Cleveland Chiropractic College Health Center, Los Angeles, California, United States
- Macquarie University, Sydney, Australia
- Durban University of Technology, Durban, South Africa